CLINICAL TRIAL: NCT00367848
Title: The Efficacy of Ultrasound in Evaluating Fractures in the Ankle and Foot in Children When the X-Ray Does Not Demonstrate Fractures.
Brief Title: Efficacy of Ultrasound in Evaluating Occult Fractures
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: SIM001- HMO-CTIL
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Fractures, Occult
Keywords: suspected fractures in the ankle and wrist
MeSH Terms: conditions — Fractures, Closed

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of the study is to examine the efficacy and accuracy of Ultrasound in evaluating occult fractures. We want to examine it on children that suffer from suspected fractures of the foot and ankle and the results of the x-ray are either negative or inconclusive.

ELIGIBILITY:
Inclusion Criteria:

* boys and girls aged <=15 years
* suspected fracture of the wrist or ankle (no later than one week after the injury)
* negative or inconclusive x-ray

Exclusion Criteria:

* unwillingness to sign informed consent

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Naum Simanovski, Dr., Principal Investigator — Hadassah Medical Organization; Natalia Simanovski, Dr., Study Chair — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel